CLINICAL TRIAL: NCT02617901
Title: COMBAT 1: COMputerised Bone Age Tool (Phase 1: Feasibility of Using Dual Energy X-ray Absorptiometry for Bone Age Assessment in Children)
Brief Title: Developing a COMputerised Bone Age Tool
Acronym: COMBAT1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SCH/14/010
Record Dates: First submitted 2015-04-23; First posted 2015-12-01 (Estimated); Results first posted 2017-10-13 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Bone Diseases, Developmental
Keywords: Bone age; Greulich & Pyle; TW3; Radiography; Dual energy x-ray absorptiometry
MeSH Terms: conditions — Bone Diseases, Developmental

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Recruited children (Experimental): Children aged below 16 years attending the Radiology Department for a left hand radiograph in order to assess bone age on the basis of clinical need. There will be one male and one female from each of five age groups (< 5 years; 5 to 7 years; 8 to 10 years; 11 to 13 years; 14 to 16 years).
  Bone age will be assessed according to the Greulich & Pyle and TW3 methods by 3 observers on 2 separate occasions at least 4 weeks apart. Recruited children will have intervention in the form of a left hand DXA which will be anonymised and from which the same 3 observers will independently assess bone age according to Greulich and Pyle and TW3 methods on 2 separate occasions at least 4 weeks apart.
  Radiographs and DXA will be read in random and varied order.
  Interventions: Radiation: Left hand DXA

INTERVENTIONS:
Radiation: Left hand DXA — All recruited children will have a left hand DXA scan which will be anonymised and from which 3 observers will independently assess bone age according to Greulich and Pyle and TW3 methods on 2 separate occasions at least 4 weeks apart.
  Radiographs and DXA will be read in random and varied order.
  Other Names: DXA of left hand and wrist

SUMMARY:
The Greulich and Pyle technique (G&P) is that most commonly used to assess bone age in children, particularly in the context of suspected skeletal dysplasia. However it has been shown not to be applicable to children of Asian and African ethnicity and may not be applicable to United Kingdom (UK) Caucasian children, who are now relatively more mature and larger than children of the mid 1930's (when G&P was developed). It is generally agreed that updated standards are required for rapid and reliable bone age assessment. The development of such standards requires irradiation of normal children. To do this ethically, radiation exposure must be kept as low as possible. Two recent studies suggest that bone age assessment can be reliably achieved from dual-energy x-ray absorptiometry (DXA) scans. As far as the investigators are aware, the Tanner & Whitehouse (TW3) method, which is preferred by some (e.g. endocrinologists and nutritionists), has not been assessed from dual-energy x-ray absorptiometry (DXA) scans - although not the main focus of this study, because of its popularity amongst certain specialties, the investigators shall be assessing the TW3 method also. Modern techniques should not only be available as textbooks, but should also be available in digital (on-line) format and where possible integrated with hospital PACS systems. The investigators believe that their team has the required experience and expertise to successfully carry out such a project. Before conducting the required large cross-sectional study, the investigators must first confirm that DXA can in fact replace radiographs for bone age assessment in children; which is the objective of this current study.

DETAILED DESCRIPTION:
This is a small prospective feasibility study to be performed over a 12-month period.

Children booked for a left hand radiograph for bone age assessment (either in isolation or as part of a dysplasia skeletal survey) will be recruited. This will require a purposive sample of 2 males and 2 females from each of the following 5 age groups (<5; 5 to 7; 8 to 10; 11 to 13; 14 to 16 years). There will therefore be a total of 20 children (10 males). Because the aim of the study is to compare results of DXA with those of radiographs in corresponding children, ethnicity of individual children will not be an issue; in other words the investigators are assessing the reliability of DXA not the reliability of G&P or TW3.

Relevant clinicians will identify patients from appropriate clinics at Sheffield Children's Hospital. Only patients having a left hand radiograph for bone age assessment on the basis of clinical need will be approached. Age appropriate information sheets will be given to them, and the study briefly discussed. When they arrive at the Radiology Department for their left hand radiograph, an appropriately certified radiographer will seek informed consent and provided the left hand radiograph is actually performed, they will then also have DXA of the left hand and those over 6 years old will be asked to complete a brief questionnaire.

Researcher 1 will anonymise hand radiographs and DXA scans, such that corresponding patient images are not identifiable. Researcher 1 will also document patient age and sex, ethnicity and body weight and height (no other clinical information is required for the purposes of this feasibility study).

Researchers 2, 3 and 4 will independently assess all images using both G&P and TW3. All observers will interpret a random selection of half the images (again independently) on a second occasion at least 2 months after the first; on both occasions the Images will be interpreted in random and varied order. Images will be read in two batches of 10 radiographs and 10 (non-corresponding) DXA scans for the first read and 5 radiographs and 5 (non-corresponding) DXA scans for the second read.

Statistical analysis is largely irrelevant for this small feasibility study. The investigators' main aim is to assess whether or not G&P and TW3 can be reliably assessed from hand DXA images.

The concordance between 1) independent readings of the three observers for radiographs and for DXA (i.e. comparing modalities) and 2) individual observers for both occasions (i.e. comparing observer reliability for each modality) will be evaluated using interclass and intraclass correlation coefficients. The investigators will calculate the mean and standard deviation of the differences between DXA and radiographs and between observers.

Statistical analyses will be performed using the Statistical Package for the Social Sciences, version 21 for Mac (SPSS, Chicago, IL).

ELIGIBILITY:
Eligibility:

1. Both female and male participants are being studied
2. Minimum age 1 year
3. Maximum age 15 years and 364 days
4. Healthy volunteers will not be recruited

Inclusion Criteria:

1. Children having a left hand radiograph performed to assess bone age on the basis of clinical need
2. Children and families who have given fully informed consent/assent
3. Children and families capable of reading and/or writing English

Exclusion Criteria:

1. Participants who might not adequately understand verbal explanations or written information given in English, or who have special communication needs

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2014-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amaka Offiah, Principal Investigator — Investigator
Locations (1):
- Sheffield Children's NHS Foundation Trust, Sheffield, Sheffield (South Yorkshire District), United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mora S, Boechat MI, Pietka E, Huang HK, Gilsanz V. Skeletal age determinations in children of European and African descent: applicability of the Greulich and Pyle standards. Pediatr Res. 2001 Nov;50(5):624-8. doi: 10.1203/00006450-200111000-00015. PMID 11641458
- [Background] van Rijn RR, Lequin MH, Robben SG, Hop WC, van Kuijk C. Is the Greulich and Pyle atlas still valid for Dutch Caucasian children today? Pediatr Radiol. 2001 Oct;31(10):748-52. doi: 10.1007/s002470100531. PMID 11685448
- [Background] Soudack M, Ben-Shlush A, Jacobson J, Raviv-Zilka L, Eshed I, Hamiel O. Bone age in the 21st century: is Greulich and Pyle's atlas accurate for Israeli children? Pediatr Radiol. 2012 Mar;42(3):343-8. doi: 10.1007/s00247-011-2302-1. Epub 2012 Jan 12. PMID 22237478

RESULTS

PARTICIPANT FLOW:
Groups:
- Recruited Children: Children aged below 16 years attending the Radiology Department for a left hand radiograph in order to assess bone age on the basis of clinical need. There was one male and one female from each of five age groups (< 5 years; 5 to 7 years; 8 to 10 years; 11 to 13 years; 14 to 16 years).
  Recruited children had intervention in the form of a left hand DXA which was anonymised and from which 2 observers independently assessed bone age according to Greulich and Pyle method on 2 separate occasions at least 4 weeks apart.
  Radiographs and DXA were read in random and varied order.
Period: Overall Study
Arm/Group | Recruited Children
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 1 male and 1 female child from each of 5 age groups as outlined in Protocol
Groups:
- Recruited Children: Children aged below 16 years attending the Radiology Department for a left hand radiograph in order to assess bone age on the basis of clinical need. There was one male and one female from each of five age groups (< 5 years; 5 to 7 years; 8 to 10 years; 11 to 13 years; 14 to 16 years).
  Recruited children had intervention in the form of a left hand DXA which was anonymised and from which the same 2 observers independently assessed bone age according to Greulich and Pyle method on 2 separate occasions at least 4 weeks apart.
  Radiographs and DXA were read in random and varied order.
Arm/Group | Recruited Children
Number analyzed (Participants) | 20
Age, Customized [Count of Participants; unit: Participants]
  Age, Customized: <5 years | 4
  Age, Customized: 5 - 7 years | 4
  Age, Customized: 8 to 10 years | 4
  Age, Customized: 11 to 13 years | 4
  Age, Customized: 14 to 16 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Region of Enrollment [Count of Participants; unit: Participants] — Children presenting to Sheffield Children's Hospital Endocrine Clinic and who required a left hand and wrist radiograph for bone age estimation.
  Participants
    United Kingdom | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Observer Agreement Between Bone Age as Assessed From Left Hand and Wrist DXA Compared to Radiographs
Description: Bone age was assessed from DXA and conventional radiographs of the left hand and wrist based on the Greulich and Pyle and Tanner and Whitehouse methods of bone age assessment.
  Interclass correlation was calculated to determine observer agreement between radiographs and DXA
Time Frame: 18 months
Population: Children presenting to Endocrine Clinic
Measure: Count of Participants; unit: Participants
Groups:
- Recruited Children: Children aged below 16 years attending the Radiology Department for a left hand radiograph in order to assess bone age on the basis of clinical need. There will be one male and one female from each of five age groups (< 5 years; 5 to 7 years; 8 to 10 years; 11 to 13 years; 14 to 16 years).
  All had left hand/wrist radiograph for bone age estimation
Arm/Group | Recruited Children
Number analyzed (Participants) | 20
Participants | 20

ADVERSE EVENTS:
Time Frame: 16 Months
Groups:
- Recruited Children: Children aged below 16 years attending the Radiology Department for a left hand radiograph in order to assess bone age on the basis of clinical need. There will be one male and one female from each of five age groups (< 5 years; 5 to 7 years; 8 to 10 years; 11 to 13 years; 14 to 16 years).
Arm/Group | Recruited Children
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No